CLINICAL TRIAL: NCT04367948
Title: Positron Nuclide Labeled NOTA-FAPI PET Study in Lymphoma
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Peking University Cancer Hospital & Institute (Other)
Responsible Party: Principal Investigator, Xuejuan Wang,MD, Principal Investigator, Peking University Cancer Hospital & Institute
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: XW-FAPI-001
Record Dates: First submitted 2020-04-26; First posted 2020-04-29 (Actual); Last update posted 2020-04-29 (Actual); Status verified 2020-04

CONDITIONS: Tumor, Solid; Positron-Emission Tomography; Lymphoma
Keywords: Lymphoma; Positron-Emission Tomography; FAPI
MeSH Terms: conditions — Neoplasms; Lymphoma

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 68Ga-NOTA-FAPI04 (Experimental): Each subject receive a single intravenous injection of 18F-FDG and 68Ga-NOTA-FAPI04, and undergo PET/CT imaging within the specified time
  Interventions: Diagnostic Test: 18F-FDG and 68Ga-NOTA-FAPI04 PET/CT
- 18F-NOTA-FAPI04 (Experimental): Each subject receive a single intravenous injection of 18F-FDG and 18F-NOTA-FAPI04, and undergo PET/CT imaging within the specified time
  Interventions: Diagnostic Test: 18F-FDG and 18F-NOTA-FAPI04 PET/CT

INTERVENTIONS:
Diagnostic Test: 18F-FDG and 68Ga-NOTA-FAPI04 PET/CT — Each subject receive a single intravenous injection of 18F-FDG and 68Ga-NOTA-FAPI04, and undergo PET/CT imaging within the specified time
  Arms: 68Ga-NOTA-FAPI04
Diagnostic Test: 18F-FDG and 18F-NOTA-FAPI04 PET/CT — Each subject receive a single intravenous injection of 18F-FDG and 18F-NOTA-FAPI04, and undergo PET/CT imaging within the specified time
  Arms: 18F-NOTA-FAPI04

SUMMARY:
To evaluate the normal physiological distribution of positron nuclide labeled NOTA-F API in human body and its detection efficiency for lymphoma

DETAILED DESCRIPTION:
Subjects first undergo an 18F-FDG test, followed by 68Ga-NOTA-FAPI04 or 18F-NOTA-FAPI04 test in groups.Investigate the standardized uptake value(SUV) of 68Ga/ 18F-NOTA-FAPI04 for the target lesion, the ratio of the standardized uptake value(SUVR) of 68Ga/ 18F-NOTA-FAPI04 for the target lesion within each time window to that of the normal corresponding tissue.

ELIGIBILITY:
Inclusion Criteria:

* ECOG score 0 or 1
* subjects with lymphoma or suspected tumor subjects who have recently (within 2 months) planned to receive pathological biopsy or tumor surgery
* expected survival ≥12 weeks
* blood routine, liver and kidney function meet the following criteria: blood routine: WBC≥4.0×109L or neutrophils ≥1.5×109L, PLT≥100×109/L, Hb≥90g/L;PT and APTT ULN 1.5 or less;Liver and kidney function: t-bil ≤1.5×ULT(upper limit of normal value), ALT/AST≤2.5ULN or ≤5×ULT(subjects with liver metastasis), ALP≤2.5ULN(ALP≤ 4.5ULN if there is bone metastasis or liver metastasis);BUN 1.5 x or less ULT, SCr 1.5 x or less ULT
* at least one measurable target lesion according to RECIST1.1
* women must use effective contraception during the study period and for 6 months after the end of the study (effective contraception means sterilization, hormone devices, condoms, contraceptives/pills, abstinence or vasectomy by a partner, etc.);Men should consent to subjects who must use contraception during the study period and for 6 months after the end of the study period
* able to understand and sign the informed consent voluntarily, with good compliance.

Exclusion Criteria:

* severe abnormalities of liver and kidney function;
* women preparing for pregnancy, pregnancy and lactation;
* cannot lie supine for half an hour;
* refuse to join the clinical researcher;
* suffering from claustrophobia or other mental illness;
* conditions that other researchers considered inappropriate for the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2020-05-01 (Estimated); Primary Completion 2021-12 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
SUV | 60 days
  Standardized uptake value of 68Ga/ 18f-nota-fapi04 for target lesion of subject or suspected tumor in each time point window (SUV)

SECONDARY OUTCOMES:
SUVR | 60 days
  the ratio of the standardized uptake value(SUVR) of 68Ga/ 18f-nota-fapi04 for the target lesion or suspected tumor lesion within each time window to that of the normal tissue corresponding to the tumor lesion or suspected tumor lesion to the standardized uptake value of 68Ga/ 18f-nota-fapi04

CONTACTS AND LOCATIONS:
Overall Officials: Zhi Yang, PhD, Study Director — Peking University Cancer Hospital & Institute
Locations (1):
- Peking University Cancer Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Chen X, Wang S, Lai Y, Wang G, Wei M, Jin X, Ding J, Zhang Y, Shi Y, Wang F, Zhu H, Yang Z, Wang X. Fibroblast Activation Protein and Glycolysis in Lymphoma Diagnosis: Comparison of 68Ga-FAPI PET/CT and 18F-FDG PET/CT. J Nucl Med. 2023 Sep;64(9):1399-1405. doi: 10.2967/jnumed.123.265530. Epub 2023 Jun 29. PMID 37385675
- [Derived] Wang G, Jin X, Zhu H, Wang S, Ding J, Zhang Y, Yang Z, Wang X. 68Ga-NOTA-FAPI-04 PET/CT in a patient with primary gastric diffuse large B cell lymphoma: comparisons with [18F] FDG PET/CT. Eur J Nucl Med Mol Imaging. 2021 Feb;48(2):647-648. doi: 10.1007/s00259-020-04946-0. Epub 2020 Jul 6. No abstract available. PMID 32632460